CLINICAL TRIAL: NCT07195747
Title: Effects of Surgical, Percutaneous or Medical Treatments for Coronary Artery Disease on Renal Function: Long-Term Outcome. Cardiorenal-trial.
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Principal Investigator, Ezio De Martino Neto, Medical Doctor (M.D.), Instituto do Coracao
Other Study IDs: 6048/25/059
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Chronic Kidney Disease
Keywords: Coronary Artery Disease; Chronic Kidney Disease; Renal Function; Coronary Artery Bypass Grafting (CABG); Percutaneous Coronary Intervention (PCI); Medical Therapy; Log-Term Outcomes
MeSH Terms: conditions — Coronary Artery Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CABG: Patients assigned to Coronary Artery Bypass Grafting (CABG)
  Interventions: Diagnostic Test: Creatinine
- PCI: Patients assigned to Percutaneous Coronary Intervention (PCI)
  Interventions: Diagnostic Test: Creatinine
- MT: Patients assigned to Medical Therapy (MT)
  Interventions: Diagnostic Test: Creatinine

INTERVENTIONS:
Diagnostic Test: Creatinine — Renal Function Follow-Up for 5 years

SUMMARY:
Background: Coronary artery disease (CAD) is treated with coronary artery bypass grafting (CABG), percutaneous coronary intervention (PCI), or optimized medical therapy (OMT). Their cardiovascular outcomes are well studied, but renal effects remain unclear.

Objective: To evaluate long-term renal outcomes of different CAD treatment strategies.

Methods: In this retrospective cohort from the MASS registry, patients with stable multivessel CAD and preserved ventricular function underwent OMT, CABG, or PCI. Annual creatinine was measured for ≥5 years, and eGFR calculated using CKD-EPI. The primary endpoint was change in renal function over time. Secondary endpoints included new-onset CKD, progression to advanced CKD, dialysis, and mortality. Analyses will use mixed-effects models and Cox regression.

Results: Over 1,700 patients met inclusion criteria. Longitudinal follow-up enables robust comparison of renal trajectories across treatment groups.

Conclusions: This trial highlights renal function as a primary outcome in CAD management, aiming to inform integrated strategies for patients with concurrent cardiovascular and renal risk.

DETAILED DESCRIPTION:
Background: Coronary artery disease (CAD) treatment strategies-coronary artery bypass grafting (CABG), percutaneous coronary intervention (PCI), or optimized medical therapy (OMT)-have well-established cardiovascular outcomes, but their long-term renal effects remain underexplored. Renal dysfunction is a key prognostic factor in CAD, yet patients with chronic kidney disease (CKD) are often underrepresented in major trials.

Objectives: To evaluate the long-term impact of surgical, percutaneous, and medical treatment strategies for stable multivessel CAD on renal function, with emphasis on estimated glomerular filtration rate (eGFR) changes and incidence of renal dysfunction.

Methods: This retrospective single-center cohort study analyzed data from the MASS registry, including patients with stable multivessel CAD, preserved left ventricular function, and baseline/annual serum creatinine measurements over ≥5 years. Eligible patients underwent OMT, CABG, or PCI (drug-eluting or bare-metal stents). Primary outcome was change in eGFR over time. Secondary outcomes included new-onset CKD (eGFR <60 mL/min/1.73 m²), progression to advanced CKD (<30 mL/min/1.73 m²), need for renal replacement therapy, and mortality. Linear mixed-effects models assessed eGFR changes; time-to-event analyses (Kaplan-Meier, Cox regression) evaluated secondary outcomes.

Results: The cohort comprised over 1,700 patients meeting inclusion criteria. Longitudinal follow-up allowed for robust assessment of renal trajectories across treatment groups. Analyses will determine whether treatment modality independently predicts renal decline, adjusting for age, sex, diabetes, hypertension, and baseline eGFR.

Conclusions: This study addresses a major evidence gap by positioning renal function as a primary outcome in CAD management. Findings may inform more integrated decision-making for patients with concurrent cardiovascular and renal risk, supporting individualized therapy selection beyond traditional cardiovascular endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Multivessel coronary artery disease (CAD) documented by angiography (2 or more epicardial arteries with stenosis of 70% or more);
* Preserved left ventricular systolic function;
* Have undergone treatment with medical therapy (MT), coronary artery bypass graft (CABG) or percutaneous coronary artery intervention (PCI), using drug-eluting stents (DES) or bare-metal stents (BMS);
* Availability of baseline serum creatinine values at the time of enrollment;
* Availability of serum creatinine measurements for a minimum of five years.

Exclusion Criteria:

* Presence of acute coronary syndrome at baseline;
* Limited life expectancy due to noncardiac comorbidities;
* Inability to maintain regular outpatient follow-up;
* Significant left main coronary artery disease (stenosis greater than 50%);
* Advanced chronic kidney disease (estimated glomerular filtration rate [eGFR] less than 30mL/min/1,73m2);
* End-stage renal disease requiring dialysis or history of kidney transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants were selected from the MASS registry, which includes individuals with angiographically confirmed CAD and regularly followed by a dedicated multidisciplinary team. Eligible patients had stable multivessel CAD and were considered suitable candidates for any of the three conventional treatment strategies: optimized medical therapy (MT), coronary artery bypass grafting (CABG), or percutaneous coronary intervention (PCI). Stable CAD was defined as ≥70% stenosis in at least two major epicardial coronary arteries, together with evidence of myocardial ischemia, either by functional stress testing or by the presence of stable angina classified as Canadian Cardiovascular Society (CCS) class I-III.
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Renal Function over Time | Over a five-year follow-up period
  The primary outcome in change in renal function over time, measured by change in eGFR

SECONDARY OUTCOMES:
Incidence of New-Onset Chronic Kidney Disease (CKD) | Over a five-year follow-up period
  Incidence of new-onset chronic kidney disease (CKD), defined as eGFR < 60mL/min/1,73m2 in patients with previously normal renal function
Progression to Advanced CKD | Over a five-year follow-up period
  Progression to advanced CKD, defined as a eGFR < 30mL/min/1,73m2
Initiation of Renal Replacement Therapy | Over a five-year follow-up period
  Initiation of renal replacement therapy, such as dialysis or kidney trnsplant
All-case mortality | Over a five-year follow-up period
Cardiovascular mortality | Over a five-year follow-up period
Cardiovascular hospitalization | Over a five-year follow-up period
  Hospitalization for heart failure or other cardiovascular events

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração (InCor) do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HCFMUSP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The datasets analyzed during the present study are available from the corresponding author upon reasonable request.